

# **Statistical Analysis Plan**

Last Updated: 30 APRIL 2022

**EPM (DCRI Only):** 8341 – RADx-UP You and Me COVID Free

#### NCT05212883

# **Investigators:**

Duke University: Michael Cohen-Wolkowiez, MD, PhD, Emily D'Agostino, DPH, Warren Kibbe, PhD, FACMI, Christoph Hornik, MD, PhD, MPH, Lisa Wruck, PhD

University of North Carolina-Chapel Hill: Giselle Corbie-Smith, MD, MSc; Gaurav Dave, MD, DrPH, MPH

Statisticians: Yang Yue, PhD; Sam Broderick, MS

Faculty Statistician: Lisa Wruck, PhD

### Table of Contents

| Background | 2 |
|------------------------------------------------|---|
| Specific Analysis Aims | |
| Study Population | |
| Intervention | |
| Outcome Variables | |
| Handling of Missing Data | |
| Analysis Objectives and Tasks | |
| APPENDIX I - Proposed Table and Figure Listing | |



### Background

The proposed project is a public health intervention with an ecological analysis component. The purpose of this public health intervention, You & Me COVID-Free (YMCF), is to mitigate the community transmission of SARS-CoV-2. This intervention contains two components. One component will be to provide thousands of households in Merced, California the opportunity to test their members frequently at home. The other component will be to promote testing and vaccination awareness and access via community-engaged strategies. CDC, NIH, and academic partners are collaborating on this public health intervention with state and local health departments, as well as community partners, to evaluate the community rollout of frequent at-home testing and the promotion of testing and vaccination awareness and access.

This study will be conducted as a non-randomized ecologic study design to assess the impact of at-home testing interventions and the promotion of vaccination in reducing community transmission in Merced County, CA. We chose Merced County based on several criteria: a) size of the population; b) proportion of Hispanic/Latino/Latinx population; c) established partnerships with the RADx-UP program and the NIH Community Engagement Alliance (CEAL); d) ongoing connection to the local health department; e) county vaccination rates; f) and county Pandemic Vulnerability Index (PVI) score. In this community, 400,000 rapid home tests obtained by the NIH have been distributed in 200,000 kits to community households. Test distribution started on Thursday, November 18, 2021, and the distribution was completed on January 22, 2022.

This cohort sub-study in a subset of the population will explore human factors in response to testing and vaccination. Participants in the public health intervention who meet eligibility criteria will be invited to participate in the sub-study, consented, and asked to complete questionnaires aimed at evaluating self-reported health conditions, COVID-19 testing and symptoms, social interactions, knowledge of prevention strategies, infection risk, and attitudes towards vaccines. This sub-study will provide participant-level information essential to understand COVID-19 testing and vaccination awareness and access and relevant for implementation of public health interventions in future pandemics.

Further details of the background and the design of the study can be found in the study proposal.

#### Specific Analysis Aims

- 1. Characterize self-reported COVID-19 testing and symptoms.
- 2. Delineate attitudes towards SARS CoV-2 vaccination.
- 3. Describe infection risk in work place.
- 4. Explore the relationship between sociodemographic factors, i.e., age, race, ethnicity, and preferred language, and
  - a. reasons for test use,
  - b. test result,
  - c. current vaccination status,
  - d. likelihood of future vaccination,
  - e. perspective on easiest way to obtain free oral COVID medicines.
- 5. Explore the relationship between social determinants of health, i.e., gender identity, employment, food/water/housing insecurity, health insurance, and COVID-19 challenges, and
  - a. testing attitude (i.e., Participant thinks it is easy to get tested for COVID-19)
  - b. testing behavior (i.e., Participant has been tested for COVID-19)



### **Study Population**

The study population will consist of people who meet the following criteria:

- Adult and child residents who are 2 years of age or greater at enrollment
- Self-report primarily residing within the intervention community (Merced County, California)
- Are participating in the public health intervention, regardless of vaccination status

The questionnaire includes three parts:

- Front Door Survey
- Baseline Survey
- End of Study Survey

A participant could scan a QR code on the participant instruction card or the You & Me COVID-Free bag to access a 1-minute Front Door Survey each time she/he takes a swab test. Individuals will also be invited to complete a more detailed Baseline Survey, which will take about 20 minutes, and then another short follow-up survey (i.e., End of Study Survey) about four weeks later. There is no consent required for each completion of the Front Door Survey and scanning the QR code will start the Front Door Survey automatically. Immediately following the Front Door Survey, the participant is asked if they would like to participate in the sub study. If they agree, they are asked to sign an informed consent form and then given the Baseline Survey to complete. The End of Study Survey is administered 28 days following the completion of the Baseline Survey. The participants who fill out the Baseline Survey and the End of Study Survey will be included in the sub study if they provide a signed and dated informed consent form. There are no exclusion criteria.

As the at-home tests are authorized for children ages 2 and up, these children may also participate in at-home testing, but they will not be enrolled as participants themselves. For children 2 to 14 years of age, an adult must collect the sample and complete the test procedure. Data will be obtained from participants at the individual level.

The Front Door Survey is administered after each swab test by scanning the QR code. There is no consent needed for the Front Door Survey. Immediately following the Front Door Survey, the Baseline Survey is administered at the time of informed consent. The End of Study Survey is administered 28 days following the completion of the Baseline Survey.

The Front Door Survey and the Baseline/End of Study Surveys cannot be linked due to the way they were set up, despite the fact that there are matching record IDs. Each entry in the Front Door Survey corresponds to a unique test result. Multiple test results can correspond to the same participant, but each test result receives a unique record ID so there is no way to link the multiple results to one participant. Each participant can sign up once to take the Baseline Survey and End of Study Survey, and each unique record ID represents one participant in the Baseline and End of Study Surveys. An observation from the Baseline and End of Study Surveys will have the same record ID as an observation in the Front Door Survey. However, this does not necessarily mean that the information across both sets of surveys are from the same participant. In order to clarify the data flow of the YMCF project, the consort diagram in Figure 1 presents data from the Front Door Survey on the number of total entries, the number of valid test results, and completeness of the primary outcomes. It also presents data from the Baseline Survey on the and number of total participants, the number of consented participants, and completeness on secondary outcomes. The primary outcomes correspond to the Front Door Survey and are:

- Participant reasons for test use
- Test result
- Current vaccination status



- Likelihood of future vaccination
- Perspective on easiest way to obtain free oral COVID medicines

Among 2,399 valid-test-result entries in Front Door Survey, 412 entries completed full set of primary outcomes, 1,987 entries partially completed primary outcomes, and none entry were missing all primary outcomes. See details in Table 1.

Table 1. Missingness of Primary Outcomes in Front Door Survey

| | Participant reasons for test use | Test<br>result | Current vaccination status | Likelihood of future vaccination | Perspective on easiest way to obtain free oral COVID medicines |
|---|---|---|---|---|---|
| Missing | 0 | 0 | 4 | 1987 | 0 |
| Not<br>missing | 2399 | 2399 | 2395 | 412 | 2399 |
| Total | 2399 | 2399 | 2399 | 2399 | 2399 |

The secondary outcomes correspond to the Baseline Survey and are:

- Participant attitudes towards SARS-CoV-2 vaccination
- Accessibility to personal protective equipment and distancing in the work place
- Self-report COVID-19 testing and symptoms

Among 1,208 consented participants in Baseline Survey, no participant completed full set of secondary outcomes, 1,208 participants partially completed secondary outcomes, and no participant were missing all secondary outcomes. See details in Table 2.

Table 2. Missingness of Secondary Outcomes in Baseline Survey

| | SARS-Co | Participant<br>attitudes towards<br>SARS-CoV-2<br>vaccination | | ssibility to personal ctive equipment and ncing in the work place | | Self-report COVID-19 testing | | Self-<br>report<br>symptoms | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Reasons<br>for<br>getting<br>COVID<br>vaccine | Reasons<br>for not<br>getting<br>COVID<br>vaccine | Have<br>access to<br>necessary<br>facilities<br>to wash | Work require to be in close contact with others | have<br>access to<br>necessary<br>personal<br>protective<br>equipment | Testing<br>method | Have<br>been<br>tested<br>for<br>COVID | Have<br>tested<br>positive<br>for<br>COVID | Accessibility to testing | 12 survey items |
| Missing | 0 | 0 | 642 | 643 | 642 | 375 | 216 | 376 | 218 | 275-381 |
| Not<br>missing | 1208 | 1208 | 566 | 565 | 566 | 833 | 992 | 832 | 990 | 827-933 |
| Total | 1208 | 1208 | 1208 | 1208 | 1208 | 1208 | 1208 | 1208 | 1208 | 1208 |



Figure 1. Consort Diagram of Front Door Survey and Baseline Survey

### **Front Door Survey**





### **Baseline Survey**



Participants for this sub-study will be recruited within Merced County, California, participating in the larger public health intervention. Recruitment strategies include marketing with public health messaging in collaboration with local health departments, community organizations, media and targeted social media outreach for awareness and education, as well as other strategies that would be tailored to the different distribution scenarios. Participants may be compensated up to \$50 for completion of all surveys. The sample size is up to 300,000 for the sub-study. The test kits distributed as part of the larger study will contain information about the sub-study and how-to consent using either a mobile application (e-consent) accessible free of charge to participants or via phone consenting (verbal consent).

All analyses will be conducted in the evaluable populations corresponding to the Front Door Survey and the Baseline Survey. The Front Door Survey Evaluable Population is defined as entries that have a valid SARS CoV-2 test response (i.e., positive or negative). The Baseline Survey Evaluable Population is defined as participants who were 2 years of age or above at enrollment, consenting to participate in the Baseline and End of Study Surveys.



#### Intervention

Test kits consisting of 2 tests per kit were distributed to Merced County households starting on November 18, 2021, through the Merced County Health Department and a coalition of community groups. Outreach and public awareness were done through a multi-pronged education and marketing program including mailers, door hangers, billboards, social media campaigns and targeted ads on local media outlets. Test kit distribution ended on December 31, 2021 and 200,000 test kits were distributed.

Text messages reminders were sent out to all study participants automatically using Twilio, with REDCap as the backend. The messages will include links to complete three surveys, i.e., Front Door Survey, Baseline Survey, and End of Study Survey (28 days later). Participant phone numbers will be provided to Twilio to facilitate the sending of text messages, and Twilio may store metadata about the delivery of the messages, such as successful or failure, and time and date stamps, but no other content will be stored. Messages for this study are one-way only and cannot be replied to.

### Outcome Variables

- Primary Outcomes (from Front Door Survey)
  - o Participant reasons for test use
  - o Participant test result
  - Participant current vaccination status
  - o Participant likelihood of future vaccination
  - o Participant perspective on easiest way to obtain free oral COVID medicines
- Secondary Outcomes (from Baseline Survey)
  - o Participant attitudes towards SARS CoV-2 vaccination
    - Proportion of reasons for getting/not getting a COVID-19 vaccination
  - o Participant accessibility to personal protective equipment and distancing in work place
    - Proportion of respondents on access to necessary personal protective and distancing
  - o Participant self-report COVID-19 testing and symptoms
    - Proportion of respondents on COVID-19 testing method, testing history and result, accessibility to testing
    - Proportion of respondents who report current symptoms

### Handling of Missing Data

No imputation will be performed for missing data. Participants who *do not know* or *prefer not to answer* a question used as an outcome variable will be treated as missing data. Survey entries which do not show a valid (positive or negative) SARS CoV-2 test result (N=111) in the Front Door Survey will not be included in the Front Door Survey Evaluable Population. Out of the 2,510 entries in the Front Door Survey, 425 completed survey items on key primary outcomes. Among the 1,313 respondents who consented to participate Baseline and End of Study Survey, 480 completed survey items on key secondary outcomes.



### Analysis Objectives and Tasks

1. **Objective:** Summarize sociodemographic characteristics and medical history of participants in the Baseline Survey Evaluable Population and summarize sociodemographic and test-relevant characteristics of entries in Front Door Survey Evaluable Population

Analysis: Sociodemographic characteristics and medical history summaries will be presented in Table 1. All the sociodemographic characteristics and medical history variables from the Baseline Survey will be summarized by age category (Adult, Minor, Overall) where Adult is defined as age ≥ 18 years of age. Similarly, sociodemographic and test-relevant characteristics of entries will be presented in Table 5. All variables are categorical and will be summarized as counts and percentages. The denominators for the percentages for each variable in Table 1 are defined as the number of participants in the Baseline Survey Evaluable Population who have non-missing data for the variable. The denominators for the percentages for each variable in Table 5 are defined as the frequency of entries in the Front Door Survey Evaluable Population which have non-missing data for the variable.

- See Appendix for proposed:
  - Table 1: Participant Sociodemographic Characteristics and Medical History in Baseline Survey in Merced County, CA
  - Table 5: Sociodemographic and Test-relevant Characteristics in Front Door Survey Entries in Merced County, CA
- **2. Objective:** Summarize self-reported COVID-19 testing characteristics and symptoms corresponding to the Baseline Survey Evaluable Population

**Analysis:** Testing method, testing history and result, accessibility to testing, and current symptoms will be presented in Table 2. All responses are taken from the Baseline Survey and will be summarized by age category (Adult, Minor, Overall). All categorical variables will be summarized as counts and percentages. The denominators for the percentages for each variable are defined as the number of participants in the Baseline Survey Evaluable Population who have non-missing data for the variable.

- See Appendix for proposed:
  - Table 2: Participant COVID-19 Testing and Symptoms in Baseline Survey in Merced County, CA
- **3. Objective:** Summarize attitudes towards SARS CoV-2 vaccination of participants in the Baseline Survey Evaluable Population

**Analysis:** Reasons for getting and not getting a COVID-19 vaccine will be presented in Table 3. All responses are taken from the Baseline Survey and will be summarized by age category (Adult, Minor, Overall). All categorical variables will be summarized as counts and percentages. The denominators for the percentages for each variable are defined as the number of participants in the Baseline Survey Evaluable Population who have non-missing data for the variable.

- See Appendix for proposed:
  - o Table 3: Participant Attitudes towards SARS CoV-2 vaccination in Baseline Survey in Merced County, CA



**4. Objective:** Summarize personal protective equipment and distancing information in the work place of participants in the Baseline Survey Evaluable Population

**Analysis:** Personal protective equipment and distancing information in work place will be presented in Table 4. All responses are taken from the Baseline Survey and will be summarized by age category (Adult, Minor, Overall). All these variables are ordinal, and they will be summarized as counts and percentages. The denominators for the percentages for each variable are defined as the number of participants in the Baseline Survey Evaluable Population who have non-missing data for the variable.

- See Appendix for proposed:
  - Table 4: Participant Infection Risk in Work Place in Baseline Survey in Merced County, CA
- **5. Objective:** Model the association between sociodemographic factors (i.e., age category, race, ethnicity, and preferred language) and the following outcomes in the Front Door Survey Evaluable Population
  - i) reasons for test use,
  - ii) test result,
  - iii) current vaccination status,
  - iv) likelihood of future vaccination.
  - v) perceived COVID-19 medication access

**Analysis:** Sociodemographic factors and outcomes will be drawn from the Front Door Survey. For the outcome i) reasons for test use, we will run a logistic regression model on each of the possible choices since participants could choose all that applied. For the outcomes ii) and iii), logistic regression will be used. For the outcome iv) likelihood of future vaccination, ordinal logistic regression will be used. For the outcome v), we will run a logistic regression model on each of the possible answers. Odds ratio estimates and 95% confidence interval will be presented in Table 6.

The methods described above will constitute the main analysis of these primary outcomes. The hypothesis is defined as:

$$H_0$$
:  $\beta_i = 0$ 

$$H_a$$
:  $\beta_i \neq 0$ 

And the logit is the linear function:  $ln(\frac{P}{1-P}) = \alpha + \beta_1 x_1 + \beta_2 x_2 + ... + \beta_k x_k$ 

Where  $\beta_i$  is the parameter coefficient of independent variable  $x_i$ , and p represents the true probability that the dependent variable y=1 (event) given the numeric values on the independent variables. This analysis will be conducted using PROC LOGISTC in SAS. The hypothesis as expressed above will be tested at a 2-sided significance level of 0.05.

Crucial assumption that must be met for logistic regression is linearity in the logit for continuous independent variables. We will use the Box-Tidwell test and scatter plot to check for linearity between the continuous predictors and the logit. If the linearity assumption is violated, it is necessary to make further adjustments either to the model (including or excluding predictors), or transforming the response and/or predictors. We will use restricted cubic splines to explore non-linear continuous associations.



It is important to note that the independence assumption for the logistic regression models may be violated since a single participant can enter multiple records in the Front Door Survey, but cannot be distinguished. If the violation is occurring then our models are underestimating standard errors, leading to inflated Type I error.

- See Appendix for proposed:
  - o Table 6: Regression estimates for the association between sociodemographic factors and COVID-19 testing, vaccination, and medication outcomes
- **6. Objective:** Model the association between social determinants of health (i.e., gender identity, employment, food/water/housing insecurity, and health insurance) and the following outcomes in the Baseline Survey Evaluable Population
  - i) testing attitude (i.e., Participant thinks it's easy to get tested for COVID-19)
  - ii) testing behavior (i.e., Participant has been tested for COVID-19)

**Analysis:** Social determinants of health and outcomes will be drawn from the Baseline Survey. For the outcome i) testing attitudes (i.e., Participant thinks it's easy to get tested for COVID-19), ordinal logistic regression will be used. For the outcome ii) testing behavior (i.e., Participant has been tested for COVID-19), logistic regression will be used. Odds ratio estimates and 95% confidence interval will be presented in Table 7.

The methods described above will constitute the main analysis of these secondary outcomes. The hypothesis is defined as:

$$H_0$$
:  $\beta_i = 0$ 

$$H_a$$
:  $\beta_i \neq 0$ 

And the logit is the linear function: 
$$\ln(\frac{P}{1-P}) = \alpha + \beta_1 x_1 + \beta_2 x_2 + \dots + \beta_k x_k$$

Where  $\beta_i$  is the parameter coefficient of independent variable  $x_i$ , and p represents the true probability that the dependent variable y=1 (event) given the numeric values on the independent variables. This analysis will be conducted using PROC LOGISTC in SAS. The hypothesis as expressed above will be tested at a 2-sided significance level of 0.05

- See Appendix for proposed:
  - o Table 7: Regression estimates for the association between social determinants of health and COVID-19 testing attitude and behavior



APPENDIX I - Proposed Table and Figure Listing



Table 1. Participant Sociodemographic Characteristics and Medical History in Baseline Survey in Merced County, CA

| Characteristic | Minor<br>(N=xxx) | Adult<br>(N=xxx) | All Respondents<br>(N=xxx) <sup>a</sup> |
|---|---|---|---|
| Age | | | |
| Median age in years | XX.X | XX.X | XX.X |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Race <sup>b</sup> | | | |
| White | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Black or African American | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| American Indian or Alaska Native | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Asian (including South Asian and Asian Indian) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Native Hawaiian or Pacific Islander | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Some other race | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Ethnicity | | | |
| Hispanic | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Gender Identify | | | |
| Woman | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Man | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Non-binary | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Transgender man | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Transgender woman | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Gender nonconforming | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Agender | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Bigender | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Current Pregnancy <sup>c</sup> | N/A | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Education | | | |



| T | | T | |
|---|---|---|---|
| Have never gone to school | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Completed 5 <sup>th</sup> grade or less | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Completed 6 <sup>th</sup> to 8 <sup>th</sup> grade | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Completed 9 <sup>th</sup> to 12 <sup>th</sup> grade | xxx (xx.x%) | xxx (xx.x%) | xxx(xx.x%) |
| Completed High school graduate or GED | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Completed Some college level/Technical/Vocational | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Completed Bachelor's degree | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Completed Master's/Doctoral degree | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Household Member | | | |
| Just me | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Living with spouse, no kids | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Family including kids | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Family with 3 generations | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Family with 4 generations | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Living with roommates | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Transitional Housing/Shelter/Homelessness | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Congregate Housing | | | |
| Group care setting | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Nursing home | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Residential care facility for disabled people | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Psychiatric treatment facility | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Group home | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Board and care home | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Prison or jail | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Halfway house | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Foster care | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Homeless or in no consistent shelter | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | · | | • • • |



| Loss of Employment due to COVID-19 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
|---|---|---|---|
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Current employment status | | | |
| Working now | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Temporarily laid off/sick leave/maternity leave | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Unemployed | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Retired | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Permanently/temporarily disabled | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Keeping house | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Student | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Essential worker | N/A | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Work place | | | |
| Nursing care facilities | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Visiting nurse/home health aide service | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Building cleaning services | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Public transportation | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Corrections facility | N/A | xxx (xx.x%) | xxx (xx.x%) |
| EMT or paramedic services | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Meat packing farm facility | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Agriculture and food production | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Grocery store | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Construction | N/A | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | N/A | xxx (xx.x%) | xxx (xx.x%) |
| Health Insurance | | | |
| No health insurance | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Private insurance | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Public insurance (Medicare/Medicaid/Tricare) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |



| Loss Health Coverage due to COVID-19 Pandemic | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
|---|---|---|---|
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Language Spoken Other than English | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Family Income | | | , |
| Less than \$15,000 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| \$15,000 - \$19,999 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| \$20,000 - \$24,999 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| \$25,000 - \$34,999 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| \$35,000 - \$49,999 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| \$50,000 - \$74,999 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| \$75,000 - \$99,999 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| \$100,000 and above | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Getting the Needed Health Care during COVID-19 | | | |
| No, not a challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes, a minor challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes, this is a major challenge | xxx (xx.x%) | xxx (xx.x%) | xxx(xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Have A Place to Stay/Live during COVID-19 | | | |
| No, not a challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes, a minor challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes, this is a major challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Getting Enough Food to Eat during COVID-19 | | | |
| No, not a challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes, a minor challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes, this is a major challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Having Clean Water to Drink during COVID-19 | | | |
| No, not a challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |



| Yes, a minor challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
|---|---|---|---|
| Yes, this is a major challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Getting the Needed Medicine during COVID-19 | | | |
| No, not a challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes, a minor challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes, this is a major challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Getting to Needed-to-Go Place during COVID-19 | | | |
| No, not a challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes, a minor challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes, this is a major challenge | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Health Conditions | | | |
| Immunocompromised condition | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Autoimmune disease | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Hypertension | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Diabetes | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Chronic kidney disease | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Cancer diagnosis and/or treatment within the past 12 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Cardiovascular disease | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Asthma | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Chronic obstructive pulmonary disease | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other chronic lung disease | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Sickle cell anemia | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Depression | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Alcohol or substance use disorder | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Intravenous drug use | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other mental health disorder | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other chronic condition | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |



- a. The total N is number of participants who consented to participate in the Baseline Survey.
- b. Participants could check all Race and Health Conditions that apply.
- c. The denominator for pregnancy is number of participants who are age 18 and beyond, biological female and also self-identify gender as woman.



Table 2. Participant COVID-19 Testing and Symptoms in Baseline Survey in Merced County, CA

| COVID-19 Testing and Symptoms | Minor<br>(N=xxx) | Adult<br>(N=xxx) | All Respondents (N=xxx) <sup>a</sup> |
|---|---|---|---|
| Able to isolate without losing job if participant tests positive for COVID-19 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Able to quarantine without losing job if participant tests positive for COVID-19 | xxx (xx.x%) | XXX (XX.X%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Participant has been tested for COVID-19 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Participant has been tested positive for COVID-19 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Month of first positive test for COVID-19 | | | |
| January | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| February | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| March | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| April | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| May | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| June | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| July | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| August | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| September | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| October | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| November | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| December | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |



| Year of first positive test for COVID-19 | | | |
|---|---|---|---|
| 2019 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| 2020 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| 2021 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| 2022 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Month of most recent test for COVID-19 | | | |
| January | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| February | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| March | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| April | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| May | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| June | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| July | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| August | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| September | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| October | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| November | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| December | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Year of most recent test for COVID-19 | | | |
| 2019 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| 2020 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| 2021 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| 2022 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Result of most recent test for COVID-19 | | | |
| Negative | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Positive | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Never obtained results | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Indeterminate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |



| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx(xx.x%) |
|---|---|---|---|
| Method of most recent test for COVID-19 | | | |
| Nasal swab | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Throat swab | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Blood sample | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Saliva | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Participant knows where to get COVID-19 testing in | | | |
| Strongly disagree | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Disagree | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Neither disagree or agree | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Agree | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Strongly agree | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Participant thinks it is easy to get tested for COVID-19 | | | |
| Strongly disagree | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Disagree | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Neither disagree or agree | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Agree | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Strongly agree | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Participant has the following symptoms during the past week | | | |
| Fever or chills | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Cough | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Shortness of breath or difficulty breathing | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Lack of energy or general tired feeling | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Muscle or body aches | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Headache | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| New loss of taste or smell | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Sore throat, congestion or runny nose | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |



| Feeling sick to your stomach or vomiting, diarrhea | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
|---|---|---|---|
| Abdominal pain | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Skin rash | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

a. The total N is number of participants who consented to participate in the Baseline Survey.



Table 3. Participant Attitudes towards SARS CoV-2 vaccination in Baseline Survey in Merced County, CA

| Vaccination Acceptance | Minor<br>(N=xxx) | Adult<br>(N=xxx) | All Respondents<br>(N=xxx) <sup>a</sup> |
|---|---|---|---|
| Participant has received a flu vaccine | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Participant has received a flu vaccine in the last 12 months | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Participant has received a COVID-19 vaccine | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Likelihood to get an approved COVID-19 vaccine when it becomes available | | | |
| Definitely not | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not at all likely | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not too likely | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Fairly likely | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Very likely | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Reason of getting a COVID-19 vaccine <sup>b</sup> | | | |
| I want to keep my family safe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I want to keep my community safe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I want to keep myself safe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I have a chronic health problem, like asthma or diabetes | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| My doctor told me to get a COVID-19 vaccine | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I don't want to get really sick from COVID-19 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I want to feel safe around other people | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I believe life won't go back to normal until most people get a COVID-19 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Required by my school or workplace | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Required for travel | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |



| Reason of NOT getting a COVID-19 vaccine <sup>c</sup> | | | |
|---|---|---|---|
| I'm allergic to vaccines | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I don't like needles | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I'm not concerned about getting really sick from COVID-19 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I'm concerned about side effects from the vaccines | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I don't think vaccines work very well | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I don't trust that the vaccines will be safe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I don't believe the COVID-19 pandemic is as bad as some people say it is | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I don't want to pay for it | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| I don't know enough about how well a COVID-19 vaccine works | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

- a. The total N is number of participants who consented to participate in the Baseline Survey.
- b. Participants could check all that apply on Reason of Getting a COVID-19 Vaccine.
- c. Participants could check all that apply on Reason of Not Getting a COVID-19 Vaccine.



Table 4. Participant Infection Risk in Work Place in Baseline Survey in Merced County, CA

| Work Place Infection Risk | Adult<br>(N=xxx) <sup>a</sup> |
|---|---|
| Participant has access to necessary facilities to wash in work place | |
| Not at all | xxx (xx.x%) |
| Rarely | xxx (xx.x%) |
| Some of the time | xxx (xx.x%) |
| Yes, most of the time | xxx (xx.x%) |
| Yes, all of the time | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) |
| Participant is in close contact (i.e. within 6 ft) with others in work place | |
| Not at all | xxx (xx.x%) |
| Rarely | xxx (xx.x%) |
| Some of the time | xxx (xx.x%) |
| Yes, most of the time | xxx (xx.x%) |
| Yes, all of the time | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) |
| Participant has access to necessary personal protective equipment in work place | |
| Not at all | xxx (xx.x%) |
| Rarely | xxx (xx.x%) |
| Some of the time | xxx (xx.x%) |
| Yes, most of the time | xxx (xx.x%) |
| Yes, all of the time | xxx (xx.x%) |
| (Missing) | xxx (xx.x%) |

a. The total N is number of participants who consented to participate in the Baseline Survey.



Table 5. Sociodemographic and Test-relevant Characteristics in Front Door Survey Entries in Merced County, CA

| Characteristic | Total Entries (N=xxx) <sup>a</sup> |
|---|---|
| Age Category <sup>b</sup> | |
| Complete survey for self | xxx (xx.x%) |
| Complete survey for child | xxx (xx.x%) |
| (missing) | xxx (xx.x%) |
| Race <sup>c</sup> | |
| White | xxx (xx.x%) |
| Black or African American | xxx (xx.x%) |
| American Indian or Alaska Native | xxx (xx.x%) |
| Asian (including South Asian and Asian Indian) | xxx (xx.x%) |
| Native Hawaiian or Pacific Islander | xxx (xx.x%) |
| Some other race | xxx (xx.x%) |
| (missing) | xxx (xx.x%) |
| Ethnicity | |
| Hispanic | xxx (xx.x%) |
| (missing) | xxx (xx.x%) |
| Main Reason for testing | |
| I wanted to be sure I/my child did not have COVID-19 before being around others | xxx (xx.x%) |
| I/my child had COVID-19 like symptoms | xxx (xx.x%) |
| I/my child was in close contact with someone who might have COVID-19 | xxx (xx.x%) |
| I/my child was in close contact with someone who tested positive for COVID-19 | xxx (xx.x%) |
| Someone in my household might have COVID-19 | xxx (xx.x%) |
| Someone in my household tested positive for COVID-19 | xxx (xx.x%) |
| Other | xxx (xx.x%) |
| (missing) | xxx (xx.x%) |
| COVID-19 test result | |
| Positive | xxx (xx.x%) |
| Negative | xxx (xx.x%) |
| (missing) | xxx (xx.x%) |



| Receive at least one dose of a COVID-19 vaccine | xxx (xx.x%) |
|---------------------------------------------------|-------------|
| (missing) | xxx (xx.x%) |
| Likelihood of future COVID-19 vaccine | |
| Very likely | xxx (xx.x%) |
| Somewhat likely | xxx (xx.x%) |
| Not very likely | xxx (xx.x%) |
| Not at all likely | xxx (xx.x%) |
| (missing) | xxx (xx.x%) |
| Easiest way to get free COVID-19 oral medications | |
| An urgent care center | xxx (xx.x%) |
| A doctor's or other health professional's office | xxx (xx.x%) |
| A mobile heath unit | xxx (xx.x%) |
| A drug store/pharmacy | xxx (xx.x%) |
| A grocery store | xxx (xx.x%) |
| A community center | xxx (xx.x%) |
| A place of worship | xxx (xx.x%) |
| A community park | xxx (xx.x%) |
| A neighborhood school | xxx (xx.x%) |
| Other | xxx (xx.x%) |
| (missing) | xxx (xx.x%) |

- a. The total entries reflect number of entries in Front Door Survey that have a valid SARS CoV-2 test response (i.e., positive or negative).
- b. Age Category is based on participant's response on the question *I am completing this survey for* each entry. If participants chose *Myself* or *Another household member* in their entries, they presumably were Adult; likewise, if *A child* were chosen in their entries, the participants presumably were children. However, there is no guarantee that *Myself* or *Another household member* is an adult, or *A child* is a child. No other valid information can be linked with Front Door Survey to identify the actual age category.
- c. Participants could check all Race that apply.



**Table 6.** Regression estimates for the association between sociodemographic factors and COVID-19 testing, vaccination, and medication outcomes

| | Reason for test use Close contact Close contact Household member COVID- 19 positive 19 positive (N= xxx) (N= xxx) (N= xxx) | | | | Positive<br>19 tes | Test result Vaccination status | | | | ire<br>ation <sup>a</sup> | Perceived easiest place to access COVID-19 oral medications Pharmacy only vs. doctor's office or community setting <sup>b</sup> (N= xxx) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| All Respondentse (N= xxx) | OR <sub>Adj</sub> <sup>c</sup> | 95% CI | OR <sub>Adj</sub> <sup>c</sup> | 95% CI | OR <sub>Adj</sub> <sup>c</sup> | 95% CI | OR <sub>Adj</sub> <sup>c</sup> | 95% CI | $OR_{Adj}^c$ | 95%<br>CI | OR <sub>Adj</sub> d | 95%<br>CI | $OR_{Adj}^{d}$ | 95% CI |
| Age, years | 3 | | , | | 3 | | 3 | | 3 | | 3 | | , | |
| <18 | x.x | X.X - X.X | x.x | x.x - x.x | X.X | X.X - X.X | x.x | x.x - x.x | X.X | X.X-<br>X.X | X.X | X.X -<br>X.X | X.X | X.X - X.X |
| ≥18 | | · | | | | • | | • | | | · | | | |
| Race | | | | | | | | | | | | | | |
| Black | x.x | X.X - X.X | X.X | X.X - X.X | X.X | x.x - x.x | X.X | X.X - X.X | X.X | X.X-<br>X.X | X.X | X.X -<br>X.X | X.X | x.x - x.x |
| Other | X.X | X.X - X.X | X.X | x.x - x.x | X.X | X.X - X.X | X.X | X.X - X.X | X.X | X.X-<br>X.X | X.X | X.X -<br>X.X | X.X | X.X - X.X |
| Asian | X.X | X.X - X.X | X.X | x.x - x.x | X.X | X.X - X.X | X.X | x.x - x.x | X.X | X.X -<br>X.X | X.X | X.X -<br>X.X | X.X | X.X - X.X |
| Multiple | X.X | X.X - X.X | X.X | X.X - X.X | X.X | X.X - X.X | X.X | X.X - X.X | X.X | X.X-<br>X.X | X.X | X.X -<br>X.X | X.X | X.X - X.X |
| White | | | | | | | | | | • | • | | | |
| Ethnicity | | | | | | | | | | | | | | |
| Hispanic/Lati<br>no/ Spanish | x.x | x.x - x.x | x.x | x.x - x.x | x.x | x.x - x.x | x.x | x.x - x.x | X.X | X.X-<br>X.X | x.x | X.X -<br>X.X | X.X | x.x - x.x |
| Non-<br>Hispanic/Lati<br>no/ Spanish | | | | | | | | | | • | | | | |



| Language | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| English | X.X | X.X - X.X | X.X | x.x - x.x | x.x | x.x - x.x | X.X | x.x - x.x | x.x | X.X-<br>X.X | X.X | X.X -<br>X.X | x.x | x.x - x.x |
| Spanish | | | | | • | | • | | • | | • | | • | |

NA=odds ratio not estimable due to small sample sizes.

Bolded estimates p<.05.

<sup>&</sup>lt;sup>a</sup>Likelihood of future vaccination per one unit change (Not at all likely to not very likely; Not very likely to somewhat likely; Somewhat likely to very likely).

<sup>&</sup>lt;sup>b</sup>Community settings=grocery store, community center, place of worship, community park, neighborhood school, or other.

<sup>&</sup>lt;sup>e</sup>Estimates based on binary logistic regression, adjusted for age, race, and ethnicity.

<sup>&</sup>lt;sup>d</sup>Estimates based ordinal logistic regression, adjusted for age, race, and ethnicity.

<sup>&</sup>lt;sup>e</sup>Number of All respondents is the number of participants who have complete data on full set of sociodemographic factors (i.e., Age, Race, Ethnicity, and Language), sample size on each outcome could vary based on the number of participants respond to the relevant survey item.



**Table 7.** Regression estimates for the association between social determinants of health and COVID-19 testing attitude and behavior in Baseline Survey

| | | ed for COVID-19 <sup>a</sup><br>= xxx) | Has been tested for COVID-19<br>(N= xxx) | |
|---|---|---|---|---|
| | | , | | , |
| All Respondents <sup>d</sup> | | | | |
| (N=xxx) | $OR_{Adj}^{b}$ | 95% CI | $OR_{Adj}{}^c$ | 95% CI |
| Gender Identify | | | | |
| Woman | X.X | X.X - X.X | X.X | X.X - X.X |
| Man | X.X | X.X - X.X | X.X | X.X - X.X |
| Non-binary | X.X | X.X - X.X | X.X | X.X - X.X |
| Transgender man | X.X | X.X - X.X | X.X | X.X - X.X |
| Transgender woman | X.X | X.X - X.X | X.X | X.X - X.X |
| Gender nonconforming | X.X | X.X - X.X | X.X | X.X - X.X |
| Agender | X.X | X.X - X.X | X.X | X.X - X.X |
| Bigender | | | • | |
| Transitional | X.X | X.X - X.X | X.X | X.X - X.X |
| Housing/Shelter/Homelessness | | | | |
| <b>Congregate Housing</b> | | | | |
| Group care setting | X.X | X.X - X.X | X.X | X.X - X.X |
| Nursing home | X.X | X.X - X.X | X.X | X.X - X.X |
| Residential care facility for | X.X | X.X - X.X | X.X | X.X - X.X |
| disabled people | | | | |
| Psychiatric treatment facility | X.X | X.X - X.X | X.X | X.X - X.X |
| Group home | X.X | X.X - X.X | X.X | X.X - X.X |
| Board and care home | X.X | X.X - X.X | X.X | X.X - X.X |
| Prison or jail | X.X | X.X - X.X | X.X | X.X - X.X |
| Halfway house | X.X | X.X - X.X | X.X | X.X - X.X |
| Foster care | X.X | X.X - X.X | X.X | X.X - X.X |
| Homeless or in no consistent | | | | |
| shelter | | | | |



| Loss of Employment due to COVID-19 | X.X | X.X - X.X | X.X | X.X - X.X |
|------------------------------------|-----|-----------|-----|-----------|
| Current employment status | | | | |
| Working now | X.X | X.X - X.X | X.X | X.X - X.X |
| Temporarily laid off/sick | | | | |
| leave/maternity leave | X.X | X.X - X.X | X.X | X.X - X.X |
| Unemployed | X.X | X.X - X.X | X.X | X.X - X.X |
| Retired | X.X | X.X - X.X | X.X | X.X - X.X |
| Permanently/temporarily | | | | |
| disabled | X.X | X.X - X.X | X.X | X.X - X.X |
| Keeping house | X.X | X.X - X.X | X.X | X.X - X.X |
| Student | X.X | x.x - x.x | X.X | X.X - X.X |
| Other | | | | |
| Health Insurance | | | | |
| No health insurance | X.X | X.X - X.X | X.X | X.X - X.X |
| Private insurance | X.X | X.X - X.X | X.X | X.X - X.X |
| Public insurance | | | | |
| (Medicare/Medicaid/Tricare) | | | | • |
| Loss Health Coverage due to | | | | |
| COVID-19 Pandemic | X.X | X.X - X.X | X.X | X.X - X.X |
| Getting the Needed Health | | | | |
| Care during COVID-19 | | | | |
| Pandemic | | | | |
| No, not a challenge | X.X | X.X - X.X | X.X | X.X - X.X |
| Yes, a minor challenge | X.X | X.X - X.X | X.X | X.X - X.X |
| Yes, this is a major challenge | | | | • |
| Have A Place to Stay/Live | | | | |
| during COVID-19 Pandemic | | | | |
| No, not a challenge | X.X | X.X - X.X | X.X | X.X - X.X |
| Yes, a minor challenge | X.X | X.X - X.X | X.X | X.X - X.X |
| Yes, this is a major challenge | • | | • | • |
| Getting Enough Food to Eat | | | | |
| during COVID-19 Pandemic | | | | |
| No, not a challenge | X.X | X.X - X.X | X.X | X.X - X.X |



| Yes, a minor challenge | X.X | x.x - x.x | X.X | x.x - x.x |
|--------------------------------|-----|-----------|-----|-----------|
| Yes, this is a major challenge | | | | |
| Having Clean Water to | | | | |
| Drink during COVID-19 | | | | |
| Pandemic | | | | |
| No, not a challenge | X.X | X.X - X.X | X.X | X.X - X.X |
| Yes, a minor challenge | X.X | X.X - X.X | X.X | X.X - X.X |
| Yes, this is a major challenge | | | | • |
| Getting the Needed Medicine | | | | |
| during COVID-19 Pandemic | | | | |
| No, not a challenge | X.X | X.X - X.X | X.X | X.X - X.X |
| Yes, a minor challenge | X.X | X.X - X.X | X.X | X.X - X.X |
| Yes, this is a major challenge | | | | |
| Getting to Needed-to-Go | | | | |
| Place during COVID-19 | | | | |
| Pandemic | | | | |
| No, not a challenge | X.X | X.X - X.X | X.X | X.X - X.X |
| Yes, a minor challenge | X.X | X.X - X.X | X.X | X.X - X.X |
| Yes, this is a major challenge | | | | |

NA=odds ratio not estimable due to small sample sizes.

Bolded estimates p<.05.

<sup>a</sup>Easy to get tested for COVID-19<sup>a</sup> per one unit change (Strongly disagree to Disagree, Disagree to Neither disagree or agree; Neither disagree or agree; Neither disagree or agree to Agee; Agree to Strongly agree).

<sup>b</sup>Estimates based on ordinal logistic regression, adjusted for gender identity.

<sup>c</sup>Estimates based on binary logistic regression, adjusted for gender identity.

<sup>d</sup>Number of All respondents is the number of participants who have complete data on full set of social determinants of health factors (i.e., gender identity, food/water/housing insecurity, employment, and health insurance), sample size on each outcome could vary based on the number of participants respond to the relevant survey item.



# **History of Changes to this Document**

| Version | Date | <b>Description of Change(s)</b> |
|---------|---------------|---------------------------------|
| 1.0 | 03 March 2022 | Initial draft |
| 2.0 | 30 April 2022 | Revision based on PIs' comments |